CLINICAL TRIAL: NCT03338556
Title: A Phase IIa, Randomised, Double-blind, Placebo-controlled Outpatients Study to Investigate the Duration of Effect and Safety of PrEP-001 Given Prophylactically in Healthy Subjects, Subsequently Challenged With Human Rhinovirus (HRV-16)
Brief Title: A Study to Examine the Duration of Effect of PrEP-001 in Healthy Subjects Challenged With HRV-16
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prep Biopharm Limited (Industry)
Collaborators: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PrEP-CS-003
Record Dates: First submitted 2017-10-20; First posted 2017-11-09 (Actual); Results first posted 2018-06-27 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Viral Upper Respiratory Tract Infection
Keywords: Rhinovirus; Healthy volunteer; Outpatient; Cold virus; HRV-16
MeSH Terms: interventions — Poly I-C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A - PrEP-001 (Active Comparator): PrEP-001 6400 μg/day, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 7 and Day - 6 prior to intranasal challenge with HRV-16 (Day 0).
  Interventions: Drug: PrEP-001
- Cohort A - Placebo (Placebo Comparator): Placebo matching PrEP-001, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 7 and Day - 6 prior to intranasal challenge with HRV-16 (Day 0).
  Interventions: Other: Placebo
- Cohort B- PrEP-001 (Active Comparator): PrEP-001 6400 μg/day, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 4 and Day - 3 prior to intranasal challenge with HRV-16 (Day 0).
  Interventions: Drug: PrEP-001
- Cohort B - Placebo (Placebo Comparator): Placebo matching PrEP-001, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 4 and Day - 3 prior to intranasal challenge with HRV-16 (Day 0).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PrEP-001
  Other Names: Poly-IC
  Arms: Cohort A - PrEP-001; Cohort B- PrEP-001
Other: Placebo
  Arms: Cohort A - Placebo; Cohort B - Placebo

SUMMARY:
A study to examine the duration of effect of PrEP-001 in healthy subjects challenged with HRV-16

DETAILED DESCRIPTION:
A phase IIa, randomised, double-blind, placebo-controlled study using outpatient setting to assess the prophylactic effect of repeated intranasal dosing of PrEP-001 in healthy subjects, subsequently challenged with HRV-16, on the changes in clinical symptoms when compared to placebo at two different dosing regimens

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 55 years on the day of first dosing with Investigational Medicinal Product (IMP).
2. In good health with no history of major medical conditions from the medical history, physical examination, and routine laboratory tests as determined by the Investigator at a screening evaluation. A subject with a history of Herpes type 1 or 2 infection may be included if there are no active lesions present and the subject is not taking active medication.
3. A total body weight ≥50 kg and Body Mass Index (BMI) ≥18 kg/m2. If the BMI is more than 30 kg/m2, the subject may be included if the waist measurement is less than 102 cm (male), or less than 88 cm (female).
4. The following inclusion criteria are applicable to subjects who are in a heterosexual relationship and female subjects in a female same sex relationship (i.e. the criteria do not apply to those in a male same sex relationship):

   1. True abstinence - when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

      Or
   2. Two forms of effective contraceptive methods among (between) the couple, which are defined as:

      • For males: i. Condom with spermicidal foam/gel/film/cream, sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. This applies only to males participating in the study).

      • For females: i. Women no longer of child bearing potential (post-menopausal females are defined as having a history of amenorrhea for at least 2 years, otherwise they should have documented status as being surgically sterile or post hysterectomy. The latter applies only to female subjects participating in the study).

      ii. If of childbearing potential, then acceptable forms of contraception include:

      o Established (a minimum of 2 weeks prior to first dosing with IMP) use of oral, injected or implanted hormonal methods of contraception.
      * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
      * Barrier methods of contraception or occlusive cap (diaphragm or cervical/vault caps), both with one of the following - spermicidal foam/gel/film/cream/suppository.

        • The longevity of contraception is as follows: i. Male subjects must comply with agreed contraception from the first IMP dosing, and continuing until 90 days after the date of the last IMP dosing or Viral Challenge which ever happens later.

      ii. Male subjects must not donate sperm following the first IMP dosing, and continuing until 90 days after the date of the last IMP dosing or Viral Challenge which ever happens later.

      iii. Female subjects of childbearing potential must have a negative pregnancy test at screening and just prior to the date of first dosing with IMP and must be using contraception consisting of two forms of birth control (one of which must be a barrier method) starting from at least 14 days prior to the first IMP dosing and continuing until 90 days after the date of the last IMP dosing or Viral Challenge whichever happens later.
5. An informed consent document signed and dated by the subject and the Investigator.
6. Sero-suitable for the Challenge Virus.
7. Subjects must be willing to comply with the protocol visit schedule including both face to face and phone visits.

Exclusion Criteria:

1. Subjects who have a significant history of any tobacco use at any time (total ≥10 pack year history [10 pack years is equivalent to one pack of 20 cigarettes a day for 10 years]).
2. Females who:

   * Are breastfeeding, or
   * Have been pregnant within 6 months prior to the study, or
   * Have a positive pregnancy test at any point during screening or prior to first dosing with IMP
3. Any history or evidence of any clinically significant cardiovascular, dermatological (including psoriasis), gastrointestinal, endocrinological, haematological, hepatic, immunological, metabolic, urological, neurological, renal, and/or other major disease that, in the opinion of the Investigator, may interfere with a subject completing the study. The following conditions apply:

   * Subjects with clinically mild atopic eczema/atopic dermatitis may be included at the Investigator's discretion (e.g., if there is no regular use of topical steroids, no eczema in cubital fossa)
   * Subjects with any history of significant psychiatric illness should be excluded unless the illness resolved within 3 months, Subjects with a diagnosis of mild or moderate depressive episode(s) which occurred 2 or more years ago, with good evidence of preceding stressors and which resolved within approximately 3 months may be included in the Investigator's opinion
   * During screening, if subjects have a total cholesterol level > 6mmol/l they will be excluded from the study.
   * Any concurrent serious illness (e.g., COPD, history of malignancy) that may interfere with a subject completing the study. Basal cell carcinoma within 5 years of initial diagnosis or with evidence of recurrence is also an exclusion
4. Abnormal pulmonary function in the opinion of the Investigator as evidenced by the responses to the respiratory screening questions and/or clinically significant abnormalities in spirometry (forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC)).
5. History or evidence of autoimmune disease or known immunodeficiency of any cause - with the exception of atopic eczema/atopic dermatitis as described in exclusion criterion number (3).
6. Subjects with any history of COPD, pulmonary hypertension, asthma or chronic lung condition of any aetiology.

   A history of childhood asthma before the age of 12 years is acceptable provided the subject is asymptomatic without treatment. Subjects with a single episode of wheezing (lasting less than 8 weeks) after age 12 years can be included at the Investigator's discretion provided the episode was more than 4 years ago and did not require a hospital admission and/or oral/intravenous steroids.
7. Positive HIV, active hepatitis A (HAV), B (HBV), or C (HCV) test.
8. Any significant abnormality altering the anatomy of the nose or nasopharynx.
9. Any clinically significant history of epistaxis (nosebleeds) within the last 12 months and/or a history of being hospitalized due to epistaxis on any previous occasion.
10. Any nasal or sinus surgery within 6 months of first dosing (due to intranasal IMP).
11. Recurrent history of fainting.
12. Twelve-lead ECG recording with clinically relevant signs of pathology and conduction disturbances as judged by the Investigator.
13. Confirmed positive test for drugs of abuse or cotinine deemed by the Investigator to be clinically significant.
14. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
15. Any clinically significant allergies such as allergy to the excipients in the Challenge Virus inoculum as stipulated in the protocol.
16. Evidence of vaccinations within the 4 weeks prior to the planned date of first dosing with IMP or an intention to receive any vaccination(s) before the last day of the study.
17. Those employed, or immediate relatives of those employed, at hVIVO or the Sponsor.
18. Receipt of blood or blood products, or loss (including blood donations) of 450 mL or more of blood during the 3 months prior to the planned date of first dosing with IMP (whichever occurs first) or planned during the 3 months after the final visit.
19. Use within 7 days prior to the planned date of first dosing with IMP of any medication or product (prescription or over-the-counter), for symptoms of hay fever, rhinitis, nasal congestion or respiratory tract infections including the use of nasal steroids.
20. Receipt of any investigational drug within 3 months prior to the planned date of first dosing with IMP or receipt of three or more investigational drugs within the previous 12 months prior to the planned date of first dosing with IMP.

    Prior inoculation with a virus from the same virus-family as the Challenge Virus or prior participation in another Human Viral Challenge study with a respiratory virus in the preceding 12 months taken from the date of first dosing with IMP in the previous study to the date of expected first dosing in this study.
21. Receipt of systemic (intravenous and/or oral) glucocorticoids or systemic antiviral drugs within 6 months prior to the planned date of first dosing with IMP. History of chemotherapy of therapy with immunomodulators.
22. History suggestive of respiratory infection within 14 days prior to first dosing or presence of significant respiratory symptoms on the day of first dosing with IMP
23. Use or anticipated use during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows, unless in the opinion of the Investigator and/or Sponsor's Medical Expert, the medication will not interfere with the study procedures or compromise subject safety. Specifically, the following are excluded:

    * Herbal supplements within 7 days prior to the planned date of first dosing with IMP
    * Chronically used medications, vitamins or dietary supplements, including any medication known to be an inducer or inhibitor of cytochrome P450 (CYP450) enzymes, within 21 days prior to the planned date of dosing with IMP
    * Over the counter medications (e.g., paracetamol or ibuprofen) where the dose taken over the preceding 7 days prior to the planned date of first dosing with IMP has exceeded the maximum permissible 24-hour dose (e.g., ≥4 g paracetamol over the preceding week)
24. Any other finding that, in the opinion of the Investigator, deems the subject unsuitable for the study.

Ages: 18 Years to 55 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Ghobadi, MD, Principal Investigator — hVIVO Services Limited
Locations (1):
- hVIVO Services Limited, QMB Innovation Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A - PrEP-001: PrEP-001 6400 μg/day, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 7 and Day - 6 prior to intranasal challenge with HRV-16 (Day 0).
  PrEP-001
- Cohort A - Placebo: Placebo matching PrEP-001, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 7 and Day - 6 prior to intranasal challenge with HRV-16 (Day 0).
  Placebo
- Cohort B- PrEP-001: PrEP-001 6400 μg/day, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 4 and Day - 3 prior to intranasal challenge with HRV-16 (Day 0).
  PrEP-001
- Cohort B - Placebo: Placebo matching PrEP-001, equally divided over both nostrils, on 2 consecutive days. Dosed Day - 4 and Day - 3 prior to intranasal challenge with HRV-16 (Day 0).
  Placebo
Period: Overall Study
Arm/Group | Cohort A - PrEP-001 | Cohort A - Placebo | Cohort B- PrEP-001 | Cohort B - Placebo
Started | 25 | 27 | 24 | 26
Completed | 23 | 23 | 22 | 24
Not Completed | 2 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - PrEP-001 | Cohort A - Placebo | Cohort B- PrEP-001 | Cohort B - Placebo | Total
Number analyzed (Participants) | 25 | 27 | 24 | 26 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 24 | 26 | 102
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (6.26) | 24.9 (8.30) | 21.7 (2.93) | 22.2 (3.58) | 23.3 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 4 | 9 | 36
  Male | 13 | 16 | 20 | 17 | 66
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 27 | 24 | 26 | 102

OUTCOME MEASURES:

1. Primary Outcome: Total Symptom Scores
Description: Overall total symptom score (TSS), defined as the sum of the total symptom scores from day 1 to day 8 inclusive, using the 10-point symptom diary card on a 0 - 3 point scale
  The following symptoms in the 10-item symptoms questionnaire were graded on a scale of 0-3, where Grade 0 was absence, Grade 1 was just noticeable, Grade 2 was bothersome but did not prevent participation in activities, and Grade 3 was bothersome and interfered with activities:
  Runny nose, Stuffy nose, Sneezing, Sore throat, Earache, Tiredness, Cough, Shortness of breath, Headache, Muscle/joint ache.
  Diary cards were filled out 3 times/day on Day 1-7 and once on Day 8. Possible range of outcomes for TSS: 0 - 660 (higher numbers indicating worse outcomes)
Time Frame: 8 days
Population: ITT analysis. Note :Cohort B PrEP-001 active group had n=21 (one less than completed the study n=22)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort A - PrEP-001 | Cohort A - Placebo | Cohort B- PrEP-001 | Cohort B - Placebo
Number analyzed (Participants) | 23 | 23 | 21 | 24
units on a scale | 22.5 (21.63) | 34.2 (38.67) | 36.2 (38.19) | 33.5 (40.54)

2. Secondary Outcome: Area Under Curve of Symptom Scores
Description: Total symptom scores (from the 10-item modified Jackson symptom diary card) were used to calculate the AUC, from Day 1 (Assessment 1) to Day 8, after challenge, for each subject using the trapezium rule, based on the available non-missing calculated total symptom scores between Day 1 (Assessment 1) and Day 8. The 10-point symptom diary card, measured three times daily was combined to generate total symptom score. The following symptoms in the 10-item symptoms questionnaire were graded on a scale of 0-3, where Grade 0 was absence, Grade 1 was just noticeable, Grade 2 was bothersome but did not prevent participation in activities, and Grade 3 was bothersome and interfered with activities:
  Runny nose, Stuffy nose, Sneezing, Sore throat, Earache, Tiredness, Cough, Shortness of breath, Headache, Muscle/joint ache
Time Frame: 8 days
Population: ITT analysis. Note :Cohort B PrEP-001 active group had n=21 (one less than completed the study n=22)
Measure: Mean (Standard Deviation); unit: scores*minutes
Arm/Group | Cohort A - PrEP-001 | Cohort A - Placebo | Cohort B- PrEP-001 | Cohort B - Placebo
Number analyzed (Participants) | 23 | 23 | 20 | 23
scores*minutes | 10668.8 (10359.03) | 16543.3 (18742.21) | 17782.2 (18533.03) | 16385.7 (19936.53)

3. Secondary Outcome: Incidence(s) of Laboratory Confirmed Illness
Description: The number of subjects with laboratory confirmed HRV-16 infection (as defined by a positive quantitative polymerase chain reaction (qPCR) result from the combined nasal washes of days 3, 4 and 5) who displayed clinical symptoms of upper respiratory tract (using the 10-item diary card, Day 1 to Day 8) - ITT analysis set
Time Frame: 8 days
Population: ITT analysis. Note :Cohort B PrEP-001 active group had n=21 (one less than completed the study n=22)
Measure: Number; unit: participants
Arm/Group | Cohort A - PrEP-001 | Cohort A - Placebo | Cohort B- PrEP-001 | Cohort B - Placebo
Number analyzed (Participants) | 23 | 23 | 21 | 24
participants | 10 | 13 | 13 | 12

ADVERSE EVENTS:
Arm/Group | Cohort A - PrEP-001 | Cohort A - Placebo | Cohort B- PrEP-001 | Cohort B - Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27 | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 19/25 | 16/27 | 18/24 | 11/26
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - PrEP-001 (N=25) | Cohort A - Placebo (N=27) | Cohort B- PrEP-001 (N=24) | Cohort B - Placebo (N=26)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 12 | 9 | 8 | 6
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 2 | 4
Blood fibrinogen increased (Investigations) | 3 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Blood and lymphatic system disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Neutropenia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nervous system disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Headache (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes